CLINICAL TRIAL: NCT03378479
Title: A Phase iv, Interventional, Non-blinded, Randomized Controlled Multicenter Study of Posaconazole Prophylaxis for the Prevention of Influenza-associated Aspergillosis (IAA) in Critically Ill Patients
Brief Title: Posaconazole for the Prevention of Influenza-associated Aspergillosis in Critically Ill Patients
Acronym: POSA-FLU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joost Wauters, prof. dr., Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POSA-FLU
Record Dates: First submitted 2017-10-30; First posted 2017-12-19 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Aspergillosis; Pulmonary, Invasive (Etiology)
Keywords: Influenza
MeSH Terms: conditions — Aspergillosis; Influenza, Human | interventions — Magnesium; posaconazole; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC + 'Posaconazole 18 MG/ML' (Other): standard of care (SOC) treatment for influenza pneumonia +posaconazole 2*300mg/d IV on day 1, followed by 1*300mg/d IV from day 2 for 7 days; vials containing 18mg posaconazole /mL, 300mg posaconazole/vial in total)
  Interventions: Drug: SOC +Posaconazole 18 MG/ML (milligram/milliliter); Other: standard of care (SOC)
- Standard of Care (Other): standard of care treatment for influenza pneumonia (at the investigators discretion)
  Interventions: Other: standard of care (SOC)

INTERVENTIONS:
Drug: SOC +Posaconazole 18 MG/ML (milligram/milliliter) — .2*300mg/d IV on day 1, followed by 1*300mg/d IV from day 2 for 7 days (total 7 days)
  Other Names: Noxafil
  Arms: SOC + 'Posaconazole 18 MG/ML'
Other: standard of care (SOC) — treatment for influenza pneumonia at the investigators discretion

SUMMARY:
The objective of this study is to deliver proof of concept that antifungal prophylaxis can reduce the incidence of Influenza Associated Aspergillosis (IAA) in ICU (intensive care unit) patients with severe influenza.

The investigators will perform an interventional non-blinded randomized controlled multicentric proof-of-concept study in patients with severe influenza admitted to the ICU. Patients will be randomized to the posaconazole prophylaxis group or to the SOC (standard of care) group. Oseltamivir will be started at the discretion of the investigator. Patients in the posaconazole group will receive posaconazole prophylaxis for 7 days.

addendum: pharmacokinetics of posaconazole as prophylaxis for invasive fungal disease on ICU

DETAILED DESCRIPTION:
Critically ill patients with PCR-confirmed influenza criteria) are eligible for inclusion in this study and will be randomized to or the posaconazole prophylaxis group or the SOC group.

If a patient is randomized to the posaconazole prophylaxis group, posaconazole (Noxafil, MSD) will be started intravenously from day 1 of randomization (2*300mg( milligram) /d on day 1, followed by 1*300mg/d from day 2 for 7 days) In both patient groups (prophylaxis and SOC) oseltamivir (non-IMP) will be started at the discretion of the treating physician from the first day of ICU admission as 2*150 mg/day for 10 days. If oseltamivir had already been started up before ICU admission, oseltamivir treatment will be continued up to a total of 10 days.

Within 48 hours after influenza diagnosis a bronchoscopy with BAL (bronchoalveolar lavage) and a serum galactomannan will be performed as part of routine ICU care in this type of patients. If an IAA-infection is suspected based on the result of this BAL ((A) Aspergillus cultured from BAL, or (B) a galactomannan (GM)the patient will be withdrawn from the study and antifungal treatment will be started.

addendum: Extensive PK sampling (UZ Leuven and Radboud): full PK curve on day 2 and day 5 (predose, 1.5; 2,3,4,6,8,10,12,18,24 h post infusion).

on non PK days, until day 7, predose sample. PK in BAL fluid only in patients with mechanical ventilation and when medically indicated.

Limited PK sampling: on day 2 and day 5: 1.5-3h, 4-8 h;8-12h; 12-24h post dose. on non PK days: PK pre dose.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the patient or his/her legal representative prior to any study procedures
2. Adult patient (≥ 18 years)
3. PCR-confirmed influenza based on nasopharyngeal swab (NS), bronchial aspirate (BA) or broncho-alveolar lavage (BAL) within 7 days before ICU admission or within 48 hours after ICU admission. If PCR is not available a positive result of a rapid test is required (a negative rapid test does not imply absence of influenza and thus requires confirmation by PCR)
4. Influenza symptoms present for no more than 10 days before ICU admission
5. Respiratory distress as the main reason for ICU admission. Respiratory distress will be defined as tachypnea with an respiratory rate ≥ 25x/min and a paO2/fiO2-ratio (fraction of inspired oxygen) ≤ 300 with or without (bilateral) infiltrates.

Exclusion Criteria:

1. Patients with age < 18 years
2. Pregnant women (based on a positive serum sample)
3. Expected survival on ICU admission ≤ 48h
4. Patients having influenza symptoms for more than 10 days before ICU admission
5. Patients being transferred from another hospital ward or another hospital who already have mycological evidence for an IAA-infection (based on sputum, BA or BAL culture, BAL or serum GM)
6. Patients with known intolerance or hypersensitivity to posaconazole or other azole antifungal agents
7. Patients that are being treated actively with antifungal agents for invasive aspergillosis
8. Patients with a QTc (corrected QT interval) interval ≥500 msec
9. Patients with liver cirrhosis (Child C)
10. Participation in another interventional clinical trial -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, Phd, Principal Investigator — UZ Leuven; Paul Verweij, Phd, Principal Investigator — Radboud University Medical Center
Locations (12):
- Belgium (4):
  - AZ Sint Jan, Bruges
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- France (3):
  - CHU Lille, Lille
  - Hospital Lariboisière, Paris
  - Hospital Saint-Louis, Paris
- Netherlands (5):
  - UMC Maastricht, Maastricht
  - UMC Radboud, Nijmegen
  - Canisius Wilhelmina Hospital, Nijmegen
  - MC Erasmus, Rotterdam
  - Elisabeth-TweeSteden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elkayal O, Mertens B, Wauters J, Debaveye Y, Rijnders B, Verweij PE, Bruggemann RJ, Spriet I, Dreesen E. Dosing of IV posaconazole to treat critically ill patients with invasive pulmonary aspergillosis: a population pharmacokinetics modelling and simulation study. J Antimicrob Chemother. 2024 Jul 1;79(7):1645-1656. doi: 10.1093/jac/dkae160. PMID 38828958
- [Derived] Vanderbeke L, Janssen NAF, Bergmans DCJJ, Bourgeois M, Buil JB, Debaveye Y, Depuydt P, Feys S, Hermans G, Hoiting O, van der Hoven B, Jacobs C, Lagrou K, Lemiale V, Lormans P, Maertens J, Meersseman P, Megarbane B, Nseir S, van Oers JAH, Reynders M, Rijnders BJA, Schouten JA, Spriet I, Thevissen K, Thille AW, Van Daele R, van de Veerdonk FL, Verweij PE, Wilmer A, Bruggemann RJM, Wauters J; Dutch-Belgian Mycosis Study Group. Posaconazole for prevention of invasive pulmonary aspergillosis in critically ill influenza patients (POSA-FLU): a randomised, open-label, proof-of-concept trial. Intensive Care Med. 2021 Jun;47(6):674-686. doi: 10.1007/s00134-021-06431-0. Epub 2021 May 29. PMID 34050768

RESULTS

PARTICIPANT FLOW:
Groups:
- SOC + 'Posaconazole 18 Milligram/Milliliter': standard of care (SOC) treatment for influenza pneumonia +posaconazole 2*300mg/d intravenously (IV) on day 1, followed by 1*300mg/d IV from day 2 for 7 days; vials containing 18mg posaconazole /mL, 300mg posaconazole/vial in total)
  SOC +Posaconazole 18 MG/ML (milligram/milliliter): .2*300mg/d IV on day 1, followed by 1*300mg/d IV from day 2 for 7 days (total 7 days)
  standard of care (SOC): treatment for influenza pneumonia at the investigators discretion
Period: Overall Study
Arm/Group | SOC + 'Posaconazole 18 Milligram/Milliliter' | Standard of Care
Started | 43 | 45
Completed | 37 | 36
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 20 | 45
  >=65 years | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (16) | 63 (15) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 23 | 18 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 37 | 36 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 4 | 5
  Belgium | 34 | 27 | 61
  France | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With IAA-infection at ICU Discharge
Description: A patient with IAA-infection is defined as a patient having mycological evidence of Aspergillus and at least one Aspergillus compatible sign or symptom and radiological abnormalities
Time Frame: from date of admission in ICU assessed up to ICU discharge, approximately 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 37 | 36
Participants | 2 | 4

2. Secondary Outcome: Time to IAPA Diagnosis
Description: Days to influenza-associated pulmonary aspergillosis (IAPA) diagnosis
Time Frame: from date of inclusion to date of first sign/symptom of IAA infection, assessed up to ICU discharge, approximately 10 days
Population: Calculated for the patients with IAPA 2 patients in SOC + 'Posaconazole 18 mg/ml' group 4 patients in SOC group
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 2 | 4
days | 10 [8 to 12] | 5 [3 to 8]

3. Secondary Outcome: Length of ICU Stay
Description: amount of days at ICU
Time Frame: from date of admission in ICU to date of discharge from ICU, approximately 20 days
Population: Length of stay was defined as the time to discharge alive, while death was considered as a competing event.
  7 patients died in SOC + POS group (37-7=30) 9 patient died in SOC group (36-9=27)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 30 | 27
days | 16 [8 to 29] | 6 [3 to 12]

4. Secondary Outcome: Length of Hospital Stay
Description: Number of days in the hospital
Time Frame: from date of admission in hospital to date of discharge from hospital, approximately 25 days
Population: Length of stay was defined as the time to discharge alive, while death was considered as a competing event.
  9 patients died in SOC + POS group (37-9=28) 11 patients died in SOC group (37-11=25)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 28 | 25
days | 25 [18 to 45] | 12 [9 to 35]

5. Secondary Outcome: ICU Mortality - Number of Participant Deaths
Description: survival status
Time Frame: At ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 37 | 36
Participants | 7 | 9

6. Secondary Outcome: Hospital Mortality - Number of Participant Deaths
Description: Survival status at hospital discharge
Time Frame: At hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 37 | 36
Participants | 8 | 10

7. Secondary Outcome: 90-day Mortality - Number of Participant Deaths
Description: Survival status at 90 days after ICU admission
Time Frame: At 90 days after ICU admission
Measure: Count of Participants; unit: Participants
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
Number analyzed (Participants) | 37 | 36
Participants | 9 | 11

ADVERSE EVENTS:
Time Frame: 90 days after ICU admission
Description: Adverse events at the ICU department are very hard to define. SAE were documented. Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | SOC + 'Posaconazole 18 MG/ML' | Standard of Care
All-Cause Mortality (participants affected / at risk) | 9/37 | 11/36
Serious Adverse Events (participants affected / at risk) | 9/37 | 11/36
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOC + 'Posaconazole 18 MG/ML' (N=37) | Standard of Care (N=36)
Death (Infections and infestations) | 9 | 11 — Not related to the study-medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOC + 'Posaconazole 18 MG/ML' (N=0) | Standard of Care (N=0)
Explanation (Infections and infestations) | NA | NA — No AEs were reported due to the ICU setting, as patients admitted to the ICU are critically ill. It is not feasible to record AEs unrelated to the study under such circumstances.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03378479/Prot_SAP_000.pdf